CLINICAL TRIAL: NCT00068991
Title: A Cluster-Randomized Trial to Evaluate the Efficacy of a Combined Individual- and Community-Based Behavioral Intervention to Improve Quality of Life for HIV-Positive Villagers in Rural China (China CIPRA Project 2)
Brief Title: HIV Educational Programs for Villagers of Funan County or Yingzhou District, Anhui Province, China
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Comprehensive International Program of Research on AIDS (Other)
Responsible Party: Rona Siskind, DAIDS
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: CIPRA Project 2; 1U19AI051915-01 (NIH); CIPRA CH 002
Record Dates: First submitted 2003-09-12; First posted 2003-09-16 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2008-09

CONDITIONS: HIV Infections
Keywords: Behavioral Intervention Study; Randomized Prevention Trial; China; Condom Use; STDs; Sexual Partners; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases | interventions — Surveys and Questionnaires; Cross-Sectional Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Participants will be HIV-infected villagers and will will take part in 2-hour skills training sessions every week from study entry to Week 8. Participants will bring a family member to each training session. After training, participants complete a post-training evaluation of the training sessions. Participants will also complete questionnaires at study entry and 6 and 12 months after completion of training.
  Interventions: Behavioral: HIV skills training program and questionnaire
- 2 (Experimental): Participants will be villagers considered influential members of their community. In the first 2 months of the study, Participants will take part in four 2-hour training sessions focusing on anti-stigma and anti-discrimination messages. Participants will also attend additional support meetings monthly, from Months 2 to 15. They will be evaluated before and after their training sessions to determine the improvements in knowledge and attitudes about HIV among group participants.
  Interventions: Behavioral: Community-level stigma reduction program
- 3 (Experimental): Participants will be randomly selected community members and will complete a cross-sectional survey at study entry and 6 and 12 months after Group 2's completion of training to determine changing community attitudes about HIV as a result of Group 2's training. There will be no additional study visits or training for Group 3 participants.
  Interventions: Behavioral: Cross-sectional survey

INTERVENTIONS:
Behavioral: HIV skills training program and questionnaire — Two-hour weekly skills training sessions followed by evaluation questionnaire
  Arms: 1
Behavioral: Community-level stigma reduction program — Two-hour training sessions focusing on anti-stigma and anti-discrimination
  Arms: 2
Behavioral: Cross-sectional survey — Survey evaluation of community attitudes towards HIV
  Arms: 3

SUMMARY:
The purpose of this study is to determine whether two educational programs about HIV will improve the quality of life of HIV infected people living in the rural villages of China. The study will enroll HIV infected adult residents, influential community members, and other community members of selected villages of Funan County or Yingzhou District, Anhui Province, China.

DETAILED DESCRIPTION:
A previous study found that HIV-infected villagers in Anhui Province, China describe their quality of life as poor. While poverty, poor health, stigma, and discrimination contribute to this poor quality of life, all these issues are interrelated and deserve further investigation. The quality of life for HIV-infected people may be made better through education, either for HIV-infected people to learn more about HIV, the treatments they are receiving, and how to deal with their disease, or for HIV uninfected people to understand HIV infection and to reduce stigma and discrimination associated with HIV infection. This study will provide skills training to HIV-infected adults and anti-stigma and anti-discrimination training to influential community members. The purpose of this study is to evaluate the changes in quality of life in HIV-infected villagers living in Anhui Province, China that result after these two training programs are administered.

There will be 3 groups in this study. Group 1 participants will be HIV-infected villagers. Group 1 participants will take part in 2-hour skills training sessions every week from study entry to Week 8. Participants will also be asked to bring a family member to each training session. After completing training, participants will be asked to complete a post-training evaluation of the training sessions. Group 1 participants will be asked to complete questionnaires at study entry and 6 and 12 months after completion of training.

Group 2 participants will be villagers considered influential members of their community. In the first 2 months of the study, Group 2 participants will take part in four, 2-hour training sessions focusing on anti-stigma and anti-discrimination messages. Group 2 participants will also attend additional support meetings monthly, from Months 2 to 15. Group 2 participants will be evaluated before and after their training sessions to determine the improvements in knowledge and attitudes about HIV among group participants.

Group 3 participants will be randomly selected community members and will complete a cross-sectional survey at study entry and 6 and 12 months after Group 2's completion of training, to determine changing community attitudes about HIV as a result of Group 2's training. There will be no additional study visits or training for Group 3 participants.

ELIGIBILITY:
Inclusion Criteria for All Participants:

* Live in one of the fourteen administrative villages in Funan County or Yingzhou District, Anhui Province, China

Inclusion Criteria for Group 1:

* HIV-infected
* Willing and able to take part in all study visits
* Willing and able to provide contact information for locator purposes
* Willing and able to bring a family member to training sessions

Inclusion Criteria for Group 2:

* Considered an influential member of their community
* Willing and able to take part in all training and follow-up support meetings

Inclusion Criteria for Group 3:

* Willing to complete the cross-sectional survey

Exclusion Criteria for All Study Participants:

* Spent more than 6 months outside of the community in the year prior to study entry
* Permanent disability (e.g., deafness, serious mental illness, mental retardation) that would interfere with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Study Completion 2007-06

PRIMARY OUTCOMES:
Medical Outcomes Study HIV Health Survey (MOS-HIV) score in-HIV infected participants | Throughout study

SECONDARY OUTCOMES:
Level of stigma among community members, as determined by HIV knowledge score and HIV attitudes and stigmatizing behaviors reported | Throughout study
Emotional well-being of HIV-infected participants, as determined by perceived support scale and stigma scale scores | Throughout study
Self-efficacy score in HIV-infected participants | Throughout study
Knowledge of correct condom use score among HIV-infected participants | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Zunyou Wu, MD, PhD, Principal Investigator — Centers for Disease Control and Prevention, China; Jie Xu, MD, MS, Principal Investigator — Centers for Disease Control and Prevention, China
Locations (1):
- Chinese Center for Disease Control and Prevention, Beijing, China